CLINICAL TRIAL: NCT07378254
Title: Co-Producing a Trauma and Substance Use Mental Health Literacy Intervention
Brief Title: Finding Emotional Empowerment and Lifelong Strength
Acronym: FEELS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alexandria Bauer, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2023000454; 1K01MH131797-01 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2026-01-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Trauma and Stressor Related Disorders; Substance Use
Keywords: mental health literacy; trauma; substance use; psychoeducation; Black and African American; young adults
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Substance-Related Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FEELS (Experimental): Finding Emotional Empowerment and Lifelong Strength
  Interventions: Behavioral: Finding Emotional Empowerment and Lifelong Strength

INTERVENTIONS:
Behavioral: Finding Emotional Empowerment and Lifelong Strength — A group-based, 12-week educational intervention to help promote mental health literacy and related beliefs, especially related to trauma and substance use.

SUMMARY:
This study will build a partnership with a Community Advisory Board to co-produce, and then pilot test, a theory-guided mental health literacy intervention focused on trauma and substance use. Participants will take part in educational group sessions for 12 weeks and complete assessments at baseline and two follow-up time points (mid-intervention and post-intervention). Intervention participants will be randomly invited to post-study focus groups to gather feedback on their experiences in the program.

DETAILED DESCRIPTION:
This study will enhance mental health literacy (i.e., knowledge and beliefs related to mental health, including recognition, prevention, and management of symptoms) among a sample of young Black adults who have experienced lifetime trauma. The culturally tailored intervention will be guided by the Theory of Planned Behavior and social ecological model as guiding frameworks. Intervention components will be designed to promote behavioral, normative, and control beliefs related to mental health care utilization, with resources to target individual, interpersonal, organizational, and community levels of influence. Following development, the intervention will be piloted among young Black adults, utilizing a single-arm pilot design.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identify as Black or African American
2. Be between the ages of 18 and 35 years old
3. Endorse previous lifetime trauma exposure
4. Participants must speak English
5. Participants are capable of giving informed consent and capable of complying with study procedures.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Multicomponent Mental Health Literacy Measure (MMHLM) | 3-months
  Assesses knowledge and beliefs about mental health disorders, including symptoms, causes, prevention and treatment strategies. Total scores range from 22 to 110, with higher scores indicating greater MHL.
Change in scores on the Short Attitudes Towards Mental Health Problems Scale (SATMHPS) | 3-months
  Measures personal, family, and community attitudes and stigma related to mental health challenges. Mean scores for subscales range from 0 to 3, with higher scores indicating more negative attitudes.
Change in scores on the Mental Help Seeking Intention Scale (MHSIS) | 3-months
  Measures intentions to seek help from a mental health professional in the event of a mental health concern. Mean scores range from from 1 to 7, with higher scores indicating stronger intentions.
Change in scores on the Self-Efficacy in Seeking Mental Health Care (SE-SMHC) | 3-months
  Assesses perceived ability to seek professional mental health care. Total scores range from 9 to 90, while subscale scores range from 5 to 50 (SE-KNOW) and 4 to 40 (SE-COPE).
Participant engagement as assessed by rates of participant recruitment and proportion of eligible participants who are enrolled in the study | 3-months
Participant satisfaction at mid- and post-intervention (quantitative) | 3-months
  Mean scores (ranging from 1 to 5) on ten Likert items assessing length of the program, pace of learning and discussing material, group format, meeting time and location, group facilitator, and program materials (i.e., amount of information given, clarity of the information given, ability to understand information, ability to apply material in real life). One additional item will ask how participants would rate the helpfulness of the FEELS intervention (1 = very unhelpful to 5 = very helpful).
Participant satisfaction at post-intervention (qualitative) | 3-months
  Three survey questions will ask participants for feedback on the intervention (facilitators for participation, topics to include in the future, and suggestions for improvement). Post-intervention focus groups will also elicit qualitative appraisals (on intervention length, pace, and modality; ease of reading, understanding, and applying the content; and suggestions for improvement) from a smaller group of intervention participants.
Participant retention and attendance at sessions | 3-months
  Mean number of intervention sessions attended per participant and proportion of participants who complete the full intervention

SECONDARY OUTCOMES:
Mental health help-seeking behaviors | 3-months
  Five questions will include looking for a mental health provider nearby, finding out whether insurance would cover a visit to a mental health provider, making an appointment, following through on the appointment, and/or visiting a provider more than once. Items will be scored as 1 = Yes and 0 = No.
Changes in scores on the Short PTSD Rating Interview (SPRINT) | 3-months
  Mean scores ranging from 0 to 4, with higher scores indicating greater PTSD symptoms.
Changes in scores on the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) | 3-months
  Mean frequency of past 3-month substance use, ranging from 0 to 6, with higher scores indicating greater substance use.

IPD SHARING:
Plan to Share IPD: No